CLINICAL TRIAL: NCT06335511
Title: Decompression Versus Instrumented Fusion for Lumbar Degenerative Disease. Clinical and Biomechanical Outcome Study
Acronym: ARCHIMEDE
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: 631-2021-OSS-AUSLBO
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Spinal Stenosis; Degenerative Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Decompression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decompression: microsurgical decompression (MiD)
  Interventions: Procedure: microsurgical decompression
- Fusion: decompression and instrumented fusion (MiD + F)
  Interventions: Procedure: decompression and instrumented fusion

INTERVENTIONS:
Procedure: microsurgical decompression — decompression of neurological structures
  Other Names: decompression
  Groups: Decompression
Procedure: decompression and instrumented fusion — decompression of neurological structures and spine stabilization
  Other Names: stabilization
  Groups: Fusion

SUMMARY:
Identification of clinical and instrumental parameters that could predict the outcome of surgical decompression of lumbar degenerative stenosis.

DETAILED DESCRIPTION:
Degenerative lumbar spine is the most common cause of chronic pain and disability with remarkable economic impact. Treatment begins with conservative options (physical combined with antalgic therapy) but often requires surgical treatment.

Two different groups of patients affected by symptomatic lumbar stenosis with no preoperative radiological signs of instability will be recruited in a prospective trial and proposed for surgery: microsurgical decompression (MiD) or decompression and instrumented fusion (MiD + F). Clinical and mechanical outcomes of two different treatments (MiD vs. MiD+F) will be compared.

An in-vitro biomechanical study will evaluate the biomechanical effect of the two surgical techniques.

The aim of this project is to obtain robust data for tailoring the surgical approach to patient individual characteristics and needs, to gain the best clinical evidence, and possibly reducing the overall costs of management of this disease.

ELIGIBILITY:
Inclusion Criteria:

* degenerative lumbar stenosis caused by bone hypertrophy, osteoarthritis of facet joints, ligamentous hypertrophy, disc protrusion
* midsagittal spinal canal diameter of 12 mm or less
* no radiological signs of instability, i.e. pathological motion on preoperative dynamic lumbar X-ray
* ongoing symptoms for a minimum of 12 weeks with no improvement to conservative treatment
* eligibility for decompression alone (MiD) or decompression and fusion (MiD+F)

Exclusion Criteria:

* congenital, traumatic, infectious and neoplastic lumbar stenosis,
* spondylolisthesis (on static X-ray), lumbar scoliosis (Cobb>10°),
* previous lumbar surgery, other types of operations (endoscopic decompression, anterior interbody fusions, interspinous devices etc.).
* patients with spine deformity requiring long fusion (i.e. >=3 levels)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (>18yrs-old) patients with symptomatic degenerative lumbar stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Short Form 12 | at baseline (day 0)
  The Short Form-12 (SF-12) healthy questionnaire is a generic standardized instrument assessing the impact of health on quality of life. It is made of twelve questions from which are calculated two different score: a Physical Component Score (with a score range 23,99 - 56,57) and a Mental Component Score (with a score range 19,06 - 60,75). The higher the number the better the outcome.
Short Form 12 | an average of 5 days (from baseline)
  The Short Form-12 (SF-12) healthy questionnaire is a generic standardized instrument assessing the impact of health on quality of life. It is made of twelve questions from which are calculated two different score: a Physical Component Score (with a score range 23,99 - 56,57) and a Mental Component Score (with a score range 19,06 - 60,75). The higher the number the better the outcome.
Short Form 12 | 1 months (day 30)
  The Short Form-12 (SF-12) healthy questionnaire is a generic standardized instrument assessing the impact of health on quality of life. It is made of twelve questions from which are calculated two different score: a Physical Component Score (with a score range 23,99 - 56,57) and a Mental Component Score (with a score range 19,06 - 60,75). The higher the number the better the outcome.
Short Form 12 | 3 months (day 90)
  The Short Form-12 (SF-12) healthy questionnaire is a generic standardized instrument assessing the impact of health on quality of life. It is made of twelve questions from which are calculated two different score: a Physical Component Score (with a score range 23,99 - 56,57) and a Mental Component Score (with a score range 19,06 - 60,75). The higher the number the better the outcome.
Visual Analogue Scale | at baseline (day 0)
  The Visual Analogue Scale (VAS) is a pain rating scale, where the minimum score is 0 (no pain) and maximum score is 10 (maximum pain imaginable).
Visual Analogue Scale | an average of 5 days (from baseline)
  The Visual Analogue Scale (VAS) is a pain rating scale, where the minimum score is 0 (no pain) and maximum score is 10 (maximum pain imaginable).
Visual Analogue Scale | 1 months (day 30)
  The Visual Analogue Scale (VAS) is a pain rating scale, where the minimum score is 0 (no pain) and maximum score is 10 (maximum pain imaginable).
Visual Analogue Scale | 3 months (day 90)
  The Visual Analogue Scale (VAS) is a pain rating scale, where the minimum score is 0 (no pain) and maximum score is 10 (maximum pain imaginable).
Oswestry Disability Index | at baseline (day 0)
  The Oswestry Disability Index (ODI) is a patient-completed questionnaire which gives a percentage score, from 0% (no disability) to 100% (complete disability), of level of function (disability). It is made of ten questions and for each question there are six possible answers.
Oswestry Disability Index | an average of 5 days (from baseline)
  The Oswestry Disability Index (ODI) is a patient-completed questionnaire which gives a percentage score, from 0% (no disability) to 100% (complete disability), of level of function (disability). It is made of ten questions and for each question there are six possible answers.
Oswestry Disability Index | 1 months (day 30)
  The Oswestry Disability Index (ODI) is a patient-completed questionnaire which gives a percentage score, from 0% (no disability) to 100% (complete disability), of level of function (disability). It is made of ten questions and for each question there are six possible answers.
Oswestry Disability Index | 3 months (day 90)
  The Oswestry Disability Index (ODI) is a patient-completed questionnaire which gives a percentage score, from 0% (no disability) to 100% (complete disability), of level of function (disability). It is made of ten questions and for each question there are six possible answers.
EuroQol-5D | at baseline (day 0)
  The EuroQol-5D (EQ-5D) is an instrument for measuring quality of life. The score is based on two part. The first part includes five questions with three answers with a range from 1 (best outcome) to 3 (worst outcome). The second part consists in a numeric scale from 0 (worst outcome) to 100 (best outcome).
EuroQol-5D | an average of 5 days (from baseline)
  The EuroQol-5D (EQ-5D) is an instrument for measuring quality of life. The score is based on two part. The first part includes five questions with three answers with a range from 1 (best outcome) to 3 (worst outcome). The second part consists in a numeric scale from 0 (worst outcome) to 100 (best outcome).
EuroQol-5D | 1 months (day 30)
  The EuroQol-5D (EQ-5D) is an instrument for measuring quality of life. The score is based on two part. The first part includes five questions with three answers with a range from 1 (best outcome) to 3 (worst outcome). The second part consists in a numeric scale from 0 (worst outcome) to 100 (best outcome).
EuroQol-5D | 3 months (day 90)
  The EuroQol-5D (EQ-5D) is an instrument for measuring quality of life. The score is based on two part. The first part includes five questions with three answers with a range from 1 (best outcome) to 3 (worst outcome). The second part consists in a numeric scale from 0 (worst outcome) to 100 (best outcome).
Postural Balance | at baseline (day 0)
  Descriptive evaluation of sway area, symmetry and visual integration performed with wearable sensors (no min or max score available).
Postural Balance | an average of 5 days (from baseline)
  Descriptive evaluation of sway area, symmetry and visual integration performed with wearable sensors (no min or max score available).
Postural Balance | 1 months (day 30)
  Descriptive evaluation of sway area, symmetry and visual integration performed with wearable sensors (no min or max score available).
Postural Balance | 3 months (day 90)
  Descriptive evaluation of sway area, symmetry and visual integration performed with wearable sensors (no min or max score available).
Locomotor performance | at baseline (day 0)
  Descriptive evaluation of similarity to reference, variability, complexity and regularity measured with wearable sensors (no min or max score available).
Locomotor performance | an average of 5 days (from baseline)
  Descriptive evaluation of similarity to reference, variability, complexity and regularity measured with wearable sensors (no min or max score available).
Locomotor performance | 1 months (day 30)
  Descriptive evaluation of similarity to reference, variability, complexity and regularity measured with wearable sensors (no min or max score available).
Locomotor performance | 3 months (day 90)
  Descriptive evaluation of similarity to reference, variability, complexity and regularity measured with wearable sensors (no min or max score available).
Spinal mobility | at baseline (day 0)
  Descriptive evaluation of spinal mobility range and smoothness measured with wearable sensors (no min or max score available).
Spinal mobility | an average of 5 days (from baseline)
  Descriptive evaluation of spinal mobility range and smoothness measured with wearable sensors (no min or max score available).
Spinal mobility | 1 months (day 30)
  Descriptive evaluation of spinal mobility range and smoothness measured with wearable sensors (no min or max score available).
Spinal mobility | 3 months (day 90)
  Descriptive evaluation of spinal mobility range and smoothness measured with wearable sensors (no min or max score available).

SECONDARY OUTCOMES:
Evaluation of costs | after 3 years
  The secondary outcome aims to compare the costs related to the two procedures themselfs (costs of the surgical procedure, hospital stay, blood transfusion, use of pain medications), but also the social costs related to absence from work (no min or max score available).

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Conti, Prof., Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna
Locations (2):
- Italy (2):
  - IRCCS Istituto Ortopedico Rizzolo, Bologna, Bologna
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Bologna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zaina F, Tomkins-Lane C, Carragee E, Negrini S. Surgical versus non-surgical treatment for lumbar spinal stenosis. Cochrane Database Syst Rev. 2016 Jan 29;2016(1):CD010264. doi: 10.1002/14651858.CD010264.pub2. PMID 26824399
- [Result] Scholler K, Alimi M, Cong GT, Christos P, Hartl R. Lumbar Spinal Stenosis Associated With Degenerative Lumbar Spondylolisthesis: A Systematic Review and Meta-analysis of Secondary Fusion Rates Following Open vs Minimally Invasive Decompression. Neurosurgery. 2017 Mar 1;80(3):355-367. doi: 10.1093/neuros/nyw091. PMID 28362963
- [Result] Ghogawala Z, Dziura J, Butler WE, Dai F, Terrin N, Magge SN, Coumans JV, Harrington JF, Amin-Hanjani S, Schwartz JS, Sonntag VK, Barker FG 2nd, Benzel EC. Laminectomy plus Fusion versus Laminectomy Alone for Lumbar Spondylolisthesis. N Engl J Med. 2016 Apr 14;374(15):1424-34. doi: 10.1056/NEJMoa1508788. PMID 27074067
- [Result] Overdevest GM, Jacobs W, Vleggeert-Lankamp C, Thome C, Gunzburg R, Peul W. Effectiveness of posterior decompression techniques compared with conventional laminectomy for lumbar stenosis. Cochrane Database Syst Rev. 2015 Mar 11;2015(3):CD010036. doi: 10.1002/14651858.CD010036.pub2. PMID 25760812
- [Result] Schmidt S, Franke J, Rauschmann M, Adelt D, Bonsanto MM, Sola S. Prospective, randomized, multicenter study with 2-year follow-up to compare the performance of decompression with and without interlaminar stabilization. J Neurosurg Spine. 2018 Apr;28(4):406-415. doi: 10.3171/2017.11.SPINE17643. Epub 2018 Jan 26. PMID 29372860
- [Result] Weiss AJ, Elixhauser A, Andrews RM. Characteristics of Operating Room Procedures in U.S. Hospitals, 2011. 2014 Feb. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #170. Available from http://www.ncbi.nlm.nih.gov/books/NBK195245/ PMID 24716251